CLINICAL TRIAL: NCT06909630
Title: Effects of Individualized PEEP Using Driving Pressure Ventilation on Postoperative Lung Complications in Robot Prostatectomy Surgery: Prospective Randomized Clinical Trial
Brief Title: Individualized PEEP and Driving Pressure Ventilation on Postoperative Lung Complications in Robot Prostatectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B-2202-737-002
Record Dates: First submitted 2023-01-11; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-06

CONDITIONS: Lung Collapse
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: In the drive group, the ventilator setting is fixed at tidal volume 6-8ml/kg and respiratory rate 15 breathes/min, and then the recruitment maneuver (RM, alveolar recruitment) is performed within the range that does not cause hemodynamic instability. After that, the PEEP is gradually raised from 5 cmH2O to 20 cmH2O. Driving pressure finds the lowest value. If there is no significant change even when the pressure change raises the PEEP, select the lowest PEEP. In the control group, PEEP is maintained in 5 cmH2O until the end of surgery.
Who Masked: Participant
Masking Description: Because a table of random numbers is used, participants do not know which group they belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): PEEP is maintained in 5 cmH2O until the end of surgery.
- Driving pressure group (Experimental): Individual PEEP is applied according to the driving pressure.
  Interventions: Other: Driving pressure group

INTERVENTIONS:
Other: Driving pressure group — individual PEEP
  Arms: Driving pressure group

SUMMARY:
In the case of robotic prostate cancer surgery under general anesthesia, the surgical posture is extreme Trendelenburg. Therefore, airway pressure is very high during mechanical ventilation, and there is a possibility of postoperative pulmonary complications. In order to prevent postoperative pulmonary complications, we tried to apply end-tidal pressure suitable for each individual to set the most tidal volume that can reduce the burden on the lungs during the perioperative period.

DETAILED DESCRIPTION:
This study is conducted on patients who are scheduled for prostate surgery under general anesthesia with robot assistance. Subjects who consented to the consent form the day before the surgery were conducted with people aged 19 years or older who belonged to the American Society of Anesthesiologists (ASA) class I or II. In the drive group, the ventilator setting is fixed at tidal volume 6-8ml/kg and respiratory rate 15 breathes/min, and then the recruitment maneuver (RM, alveolar recruitment) is performed within the range that does not cause hemodynamic instability. After that, the PEEP is gradually raised from 5 cmH2O to 20 cmH2O. Driving pressure finds the lowest value. If there is no significant change even when the pressure change raises the PEEP, select the lowest PEEP. In the control group, PEEP is maintained in 5 cmH2O until the end of surgery. The primary outcome of the study is to confirm the presence or absence of postoperative pulmonary complications using Chest X-rays, vital signs, and blood tests. It is the individualized PEEP value as a secondary outcome. The related driving pressure and compliance will also be observed. In addition, anesthesia/surgical time, use of vasopressors, amount of blood loss, amount of fluid, and amount of urine will be measured.

ELIGIBILITY:
Inclusion Criteria:

* elective RALP surgery under genenal anesthesia
* ASA 1-2
* 19 years of age or older
* Consented to participate in the study

Exclusion Criteria:

* Do not consent to participate in the study
* ≥ BMI 40 kg/m2
* Moderate or severe obstructive/restrictive pulmonary disease on pulmonary function tests
* Preoperative serious cardiovascular disease
* Required postoperative ventilator care at ICU care

Ages: 19 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Post operative pulmonary complication(PPC) | up to PostOperative Day(POD) #3
  Post operative lung complication

SECONDARY OUTCOMES:
Individual ventilatory setting | during opertaion
  PEEP in cmH2O at mechanical ventilation setting static lung compliance in liters/cmH2O at measured mechanical ventilation and calculated driving pressure in cmH20 Driving pressure (DP or ΔP) is defined as the distending pressure above the applied positive end-expiratory pressure (PEEP) required to generate tidal volume (VT)
  * C stat= tidal volume/ Driving pressure
  * Driving pressure= tidal volume/C stat
blood pressure(hypotension) | during opertaion
  Types and dosages of vasopressor agents used when the mean blood pressure is ≤ 60 mmHg.
  ** vasopressor agents: Ephedrine, phenylepherine, Norepinepherine
  * Ephedrine single intravenous injection: 5mg
  * phenylepherine single intravenous injection: 20mcg continueous infusion: mcg/kg/min at 100mcg/cc
  * Norepinepherine continueous infusion: mcg/kg/min at 10mcg/cc

CONTACTS AND LOCATIONS:
Overall Officials: Yu kyung Bae, Principal Investigator — SNUBH
Locations (1):
- SNUBH, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No